CLINICAL TRIAL: NCT01222091
Title: Effect of Beta Blockade on Opioid-Induced Hyperalgesia in Humans
Brief Title: Study on the Effect of a Beta Blocker on Increased Sensitivity to Pain in Humans Caused by Opioids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Larry Fu-nien Chu, Professor of Anesthesia, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SU-10062010-7050
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Results first posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-05

CONDITIONS: Hyperalgesia
MeSH Terms: conditions — Hyperalgesia | interventions — Propranolol; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propranolol, Then Placebo (Active Comparator): Propranolol, a beta blocker, or placebo to match, will be given to test whether or not it could modulate the expression of remifentanil-induced postinfusion hyperalgesia (RPH) during two pain test including: mechanically evoked pain to map the size of the hyperalgesic skin region caused by electrical stimulation and heat pain.
  Interventions: Drug: Propranolol; Drug: Placebo to Match Propranolol; Drug: Remifentanil
- Placebo, Then Propranolol (Placebo Comparator): Propranolol, a beta blocker, or placebo to match, will be given to test whether or not it could modulate the expression of remifentanil-induced postinfusion hyperalgesia (RPH) during two pain test including: mechanically evoked pain to map the size of the hyperalgesic skin region caused by electrical stimulation and heat pain.
  Interventions: Drug: Propranolol; Drug: Placebo to Match Propranolol; Drug: Remifentanil

INTERVENTIONS:
Drug: Propranolol — Propranolol administered intravenously, initially set to target plasma concentration of 5 ng/mL, titrated upward in 5 ng/mL intervals until a final concentration of 15 ng/mL is achieved.
  Other Names: Hemangeol; Inderal; Innopran
Drug: Placebo to Match Propranolol
Drug: Remifentanil — Remifentanil administered intravenously at a plasma concentration of 3 ng/mL.

SUMMARY:
This research study explores whether a beta-blocker (propranolol) can prevent a person from becoming more sensitive to pain after administration of an opioid (remifentanil). Beta blockers inhibit the sympathetic (fight or flight) response and are often used to treat angina and high blood pressure. In a previous study in human volunteers, the investigators demonstrated an increased sensitivity to pain after a 60-minute infusion of the opioid remifentanil. The goal of this study is to identify a possible inhibitor of this phenomenon.

DETAILED DESCRIPTION:
Recent evidence suggests that opioid therapy may cause a biphasic response, i.e. initial pain relief followed paradoxically by a longer lasting hypersensitivity to pain. Recent genetic analysis in mice suggests that beta adrenergic receptor antagonists reduce opiate-induced hyperalgesia (OIH). The purpose of this study is to determine the analgesic and antihyperalgesic properties of the beta-blocker propranolol on remifentanil-induced hypersensitivity in humans.

The investigators want to determine the analgesic and antihyperalgesic properties of the beta-blocker propranolol on remifentanil-induced hypersensitivity in humans. The investigators hope to learn whether the administration of beta-blocker propranolol will significantly diminish the hyperalgesic response after administration of an opioid.

The primary outcome measure for this study is change in size (area) of secondary hyperalgesia after cessation of remifentanil infusion, a measure of OIH.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men,
2. Age between 18 and 45 years
3. Normal weight (according to the table provided by Metropolitan Life Insurance).

Exclusion Criteria:

1. Hypersensitivity to opioids or naloxone,
2. History of addictive disease,
3. Significant cardiac, respiratory, gastrointestinal, neurological, dermatological, and psychiatric diseases,
4. Concurrent medication with an analgesic drug,
5. Student and employees affiliated with our laboratory

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-02; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Larry Fu-nien Chu, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chia YY, Liu K, Wang JJ, Kuo MC, Ho ST. Intraoperative high dose fentanyl induces postoperative fentanyl tolerance. Can J Anaesth. 1999 Sep;46(9):872-7. doi: 10.1007/BF03012978. PMID 10490157
- [Background] Guignard B, Bossard AE, Coste C, Sessler DI, Lebrault C, Alfonsi P, Fletcher D, Chauvin M. Acute opioid tolerance: intraoperative remifentanil increases postoperative pain and morphine requirement. Anesthesiology. 2000 Aug;93(2):409-17. doi: 10.1097/00000542-200008000-00019. PMID 10910490
- [Background] Larcher A, Laulin JP, Celerier E, Le Moal M, Simonnet G. Acute tolerance associated with a single opiate administration: involvement of N-methyl-D-aspartate-dependent pain facilitatory systems. Neuroscience. 1998 May;84(2):583-9. doi: 10.1016/s0306-4522(97)00556-3. PMID 9539228
- [Background] Laulin JP, Larcher A, Celerier E, Le Moal M, Simonnet G. Long-lasting increased pain sensitivity in rat following exposure to heroin for the first time. Eur J Neurosci. 1998 Feb;10(2):782-5. doi: 10.1046/j.1460-9568.1998.00083.x. PMID 9749743
- [Background] Laulin JP, Maurette P, Corcuff JB, Rivat C, Chauvin M, Simonnet G. The role of ketamine in preventing fentanyl-induced hyperalgesia and subsequent acute morphine tolerance. Anesth Analg. 2002 May;94(5):1263-9, table of contents. doi: 10.1097/00000539-200205000-00040. PMID 11973202
- [Background] Li X, Angst MS, Clark JD. Opioid-induced hyperalgesia and incisional pain. Anesth Analg. 2001 Jul;93(1):204-9. doi: 10.1097/00000539-200107000-00040. PMID 11429366
- [Background] Celerier E, Laulin JP, Corcuff JB, Le Moal M, Simonnet G. Progressive enhancement of delayed hyperalgesia induced by repeated heroin administration: a sensitization process. J Neurosci. 2001 Jun 1;21(11):4074-80. doi: 10.1523/JNEUROSCI.21-11-04074.2001. PMID 11356895
- [Background] Compton P, Charuvastra VC, Kintaudi K, Ling W. Pain responses in methadone-maintained opioid abusers. J Pain Symptom Manage. 2000 Oct;20(4):237-45. doi: 10.1016/s0885-3924(00)00191-3. PMID 11027904
- [Background] Liang DY, Liao G, Wang J, Usuka J, Guo Y, Peltz G, Clark JD. A genetic analysis of opioid-induced hyperalgesia in mice. Anesthesiology. 2006 May;104(5):1054-62. doi: 10.1097/00000542-200605000-00023. PMID 16645459
- [Background] Troster A, Sittl R, Singler B, Schmelz M, Schuttler J, Koppert W. Modulation of remifentanil-induced analgesia and postinfusion hyperalgesia by parecoxib in humans. Anesthesiology. 2006 Nov;105(5):1016-23. doi: 10.1097/00000542-200611000-00024. PMID 17065897
- [Background] Shafer SL, Varvel JR, Aziz N, Scott JC. Pharmacokinetics of fentanyl administered by computer-controlled infusion pump. Anesthesiology. 1990 Dec;73(6):1091-102. doi: 10.1097/00000542-199012000-00005. PMID 2248388
- [Background] Drover DR, Lemmens HJ. Population pharmacodynamics and pharmacokinetics of remifentanil as a supplement to nitrous oxide anesthesia for elective abdominal surgery. Anesthesiology. 1998 Oct;89(4):869-77. doi: 10.1097/00000542-199810000-00011. PMID 9778004
- [Background] Schmelz M, Schmid R, Handwerker HO, Torebjork HE. Encoding of burning pain from capsaicin-treated human skin in two categories of unmyelinated nerve fibres. Brain. 2000 Mar;123 Pt 3:560-71. doi: 10.1093/brain/123.3.560. PMID 10686178
- [Background] Koppert W, Dern SK, Sittl R, Albrecht S, Schuttler J, Schmelz M. A new model of electrically evoked pain and hyperalgesia in human skin: the effects of intravenous alfentanil, S(+)-ketamine, and lidocaine. Anesthesiology. 2001 Aug;95(2):395-402. doi: 10.1097/00000542-200108000-00022. PMID 11506112
- [Background] Avram MJ, Krejcie TC, Henthorn TK, Niemann CU. Beta-adrenergic blockade affects initial drug distribution due to decreased cardiac output and altered blood flow distribution. J Pharmacol Exp Ther. 2004 Nov;311(2):617-24. doi: 10.1124/jpet.104.070094. Epub 2004 Jun 14. PMID 15197245
- [Result] Chu LF, Cun T, Ngai LK, Kim JE, Zamora AK, Young CA, Angst MS, Clark DJ. Modulation of remifentanil-induced postinfusion hyperalgesia by the beta-blocker propranolol in humans. Pain. 2012 May;153(5):974-981. doi: 10.1016/j.pain.2012.01.014. Epub 2012 Feb 22. PMID 22365565

RESULTS

PARTICIPANT FLOW:
Groups:
- Propranolol, Then Placebo: Half of the participants received propranolol at the first study session and the saline placebo at the second session. The treatment infusions were administered continuously before, during, and after remifentanil infusion.
- Placebo, Then Propranolol: Half of the participants received saline placebo at the first study session and propranolol at the second session. The treatment infusions were administered continuously before, during, and after remifentanil infusion.
Period: Overall Study
Arm/Group | Propranolol, Then Placebo | Placebo, Then Propranolol
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Half of the participants received propranolol at the first study session and the saline placebo at the second session. The treatment infusions were administered continuously before, during, and after remifentanil infusion.
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 23.8 [18 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Weight [Mean (Full Range); unit: kilograms] | 78.8 [57 to 130]
Height [Mean (Full Range); unit: centimeters] | 178 [168 to 194]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Size (Area) of Secondary Hyperalgesia After Cessation of Remifentanil Infusion, a Measure of Opioid-induced Hyperalgesia (OIH).
Description: A slightly modified version of a previously described model of secondary hyperalgesia was used. Two copper wires contained in a microdialysis catheter were inserted in parallel over a length of 5 mm into the dermis of the right volar forearm. The wires were connected to a constant current stimulator controlled by a pulse generator to deliver rectangular and monophasic pulses with a duration of 0.5 mg at 2 Hz. Over a period of 15 min, the current was increased by targeting a pain rating of 5 on an 11-point numeric rating scale (0 = no pain and 10 = maximum tolerable pain) until the hyperalgesic area surrounding the stimulation site was fully established. Once the area was established, the current was held constant. Percent change from baseline in size (area) of secondary hyperalgesia after cessation of remifentanil infusion was calculated per group.
Time Frame: Baseline; 15 min post remifentanil (REM) infusion; 60 min post REM infusion
Measure: Number; unit: percentage of change
Groups:
- Propranolol; Placebo: Half of the participants received propranolol at the first study session and the saline placebo at the second session. The treatment infusions were administered continuously before, during, and after remifentanil infusion.
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 10 | 10
percentage of change
  15 min post remifentanil infusion | -28 | -34
  60 min post remifentanil infusion | -19 | 141.5

2. Secondary Outcome: Objective Opioid Withdrawal Scale (OOWS)
Description: OOWS: Is a 13-item instrument of documenting physically observable signs of withdrawal, which are rated as present (1) or absent (0) during the observation period. Maximum score = 13, minimum score = 0. Lower scores correspond to fewer symptoms.
Time Frame: Pretreatment [90 min prior to 60-min REM infusion]; 30 min prior to 60-min REM infusion; 15 and 40 min after start of 60-min REM infusion; 5, 15, and 75 minutes after finish of 60-min REM infusion)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 10 | 10
units on a scale
  Pretreatment | 1.2 (1.5) | 1.1 (1.3)
  30 min prior to REM infusion | 1.1 (2) | 1.1 (1)
  15 min after start of REM infusion | 0.1 (2) | 0.8 (1)
  40 min after start of REM infusion | 0.8 (2) | 0.5 (1)
  5 minutes after finish of REM infusion | 3 (4) | 1.8 (2)
  15 minutes after finish of REM infusion | 2.8 (4.2) | 2.1 (2.1)
  75 minutes after finish of REM infusion | 1.7 (4) | 1.6 (2)

ADVERSE EVENTS:
Arm/Group | Propranolol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Local anesthetic properties of propranolol; electrical burn pain model not useful for fully reproducing clinical sources of pain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No